CLINICAL TRIAL: NCT05503342
Title: Pharmacotherapy Follow-up of a Randomized Cohort to Monitor Patients With Asthma on Well-defined Treatment Using a Self-management Mobile Application
Brief Title: Monitoring of Patients With Asthma Performed by a Clinical Pharmacist Using a Mobile Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rafael Stelmach (Other)
Collaborators: Federal University of Amazonas (Other)
Responsible Party: Sponsor-Investigator, Rafael Stelmach, Collaborating Professor, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SDC - 4874/19/093
Record Dates: First submitted 2022-08-10; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Asthma
Keywords: Asthma; Pharmaceutical Services; Pharmacists; Self-Management; Mobile Applications
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: In both arms, patients will be followed up in a 12-week pharmacotherapeutic follow-up program, where they will have to record weekly three measurements of peak expiratory flow and fill out a questionnaire to assess the control on paper (control group) or fill out a risk score for exacerbation contemplated in the mobile application, which the pharmacist will have access through a web platform (intervention group). Depending on the evolution of each patient, the pharmacist will provide the relevant guidelines to improve control, as well as referral to a medical care service, if applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): They will be followed up in a 12-week pharmacotherapeutic follow-up program, where they will have to record three measurements of peak expiratory flow weekly and fill out a questionnaire to assess control on paper.
  Depending on the evolution of each patient, the pharmacist will provide the relevant guidelines to improve control, as well as referral to a medical care service, if applicable.
  Interventions: Other: Asthma control assessment
- Application (Experimental): They will be followed up in a 12-week pharmacotherapeutic follow-up program, where they will have to record three measurements of peak expiratory flow weekly and fill in an exacerbation risk score included in the cell phone application, which the pharmacist will have access to through a web platform. Depending on the evolution of each patient, the pharmacist will provide the relevant guidelines to improve control, as well as referral to a medical care service, if applicable.
  Interventions: Other: Mobile Application

INTERVENTIONS:
Other: Mobile Application — Use of the cell phone application to include information about asthma symptoms which had returned with guidance on self-management.
  Arms: Application
Other: Asthma control assessment — Asthma control assessment questionnaire application in paper format
  Arms: Control

SUMMARY:
Asthma is a chronic inflammatory disease that affects the lungs. In Brazil it is responsible for about 4 to 8 deaths per day. Pharmacotherapeutic follow-up programs for people with asthma have a positive impact on treatment adherence, as well as on education about the disease, helping patients in their self-management and recognition of their health status. The use of mobile applications that assist in the monitoring and self-management of people with asthma has been increasing significantly, but we do not have much information about their real impact on the control of the disease. Thus, the aim of this study is to evaluate the use of a mobile application in the monitoring and self-management of symptoms in adults with asthma in a pharmaceutical care program at a university outpatient clinic in São Paulo, Brazil.

DETAILED DESCRIPTION:
Study design: interventional study

Patients will be selected according to eligibility criteria and after having agreed and signed an informed consent form, they will be randomized into one of the arms of the study.

At the inclusion visit, demographic data, health history, medication history and allergy history will be collected. They will be evaluated regarding the level of asthma control using the ACQ-6 instrument, as well as the ability to use inhaled medications. They will receive the relevant guidelines regarding the activities that will be carried out during the study.

In both arms, patients will be followed up in a 12-week pharmacotherapeutic follow-up program, where they will have to record weekly three measurements of peak expiratory flow and fill out a questionnaire to assess the control on paper (control group) or fill out a risk score for exacerbation contemplated in the mobile application, which the pharmacist will have access through a web platform (intervention group). Depending on the evolution of each patient, the pharmacist will provide the relevant guidelines to improve control, as well as referral to a medical care service, if applicable.

During the study, a follow-up visit will be carried out and, at the end of the 12 weeks, a closing visit, where will be evaluated the need for medical support during the period, the use of systemic corticosteroids, access to control treatment, the occurrence of adverse event, review of pharmacotherapy and inhalation technique.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of asthma and being under medical follow-up for at least six months;
* Meet at least one of the following criteria: a) Have had at least one (01) exacerbation in the last 12 months; b) Have used oral corticosteroids in the last three months; and/or c) Being using high doses of inhaled corticosteroid (budesonide > 800 mcg/day; fluticasone > 500 mcg/day; or beclomethasone > 400 mcg/day - pressurized HFA gas-based device or >1000 mcg/day - other devices).
* Understand, agree and sign the Free and Informed Consent Term.

Exclusion Criteria:

* Illiterate patients or patients with cognitive deficits;
* Patients not fluent in Portuguese;
* Patients without mobile device skills;
* Patients who do not have mobile devices with Android® 6.0 operating system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2022-04-23 (Actual); Study Completion 2022-04-23 (Actual)

PRIMARY OUTCOMES:
Change in Asthma Control at 4 weeks | 4 weeks after the inclusion visit
  The evolution of asthma control will be evaluated through repeated measures of a validated control assessment questionnaire (control arm) or by the risk of exacerbation score contemplated in the cell phone application (application arm)
Change in Asthma Control at 12 weeks | 12 weeks after the inclusion visit
  The evolution of asthma control will be evaluated through repeated measures of a validated control assessment questionnaire (control arm) or by the risk of exacerbation score contemplated in the cell phone application (application arm)
Occurrence of exacerbations | Up to study completion, an average of 12 weeks
  Assessment of the number of occurrences of severe exacerbations that required medical support.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Stelmach, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Hospital das Clincias da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No